CLINICAL TRIAL: NCT01869426
Title: Impact of VSL#3 on Infants Colics as Assessed by Average Crying Time
Brief Title: Impact of Probiotic Preparation VSL#3 on Infants Colics
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Prof. Maria Elisabetta Baldassarre, Professor of Pediatrics, Policlinico Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VSLcolics13
Record Dates: First submitted 2013-05-28; First posted 2013-06-05 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Infant Colics
Keywords: colics
MeSH Terms: conditions — Colic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VSL#3 drops (Active Comparator): 31 infants will receive 10 drops active product that should be taken daily (preferably in the morning before feeding) for 21 days.
  Interventions: Dietary Supplement: VSL#3 drops
- VSL#3 drops placebo (Placebo Comparator): 31 infants will receive 10 drops of placebo product that should be taken daily (preferably in the morning before feeding) for 21 days.
  Interventions: Dietary Supplement: VSL#3 drops placebo

INTERVENTIONS:
Dietary Supplement: VSL#3 drops
  Arms: VSL#3 drops
Dietary Supplement: VSL#3 drops placebo
  Arms: VSL#3 drops placebo

SUMMARY:
Infantile colic is one of the most commonly reported medical problems within the first three months of life causing appreciable distress for both parents and pediatricians.

It appears that multiple independent origins might be involved: amongst them infant's difficult temperament, inadequate mother-infant communication or maternal anxiety, transient lactase deficiency, exposure to cow's milk, abnormal gastrointestinal function, maternal smoking during pregnancy or after delivery. Consequently, various treatment approaches have been tried to alleviate this condition.

Recent studies have suggested that changes of intestinal microflora of a newborn may play an important role in pathogenesis of infantile colic. Therefore, dietary supplementation with probiotics has been proposed for the improvement of this condition.

DETAILED DESCRIPTION:
Aim of the study is to evaluate the improvement of colics symptoms by the oral administration of VSL#3 and the difference in the daily average crying time (measured with parental diary) between end of treatment and baseline.

In this study, 62 infants will be enrolled and will receive 10 drops per day of VSL#3 or Placebo according to randomization list. The study product will be supplied as a box containing the oil bottle and a powder stick. The product should be stored refrigerated. On the first day of supplementation, the mother will open the sachet, pour the contents into the bottle and shake vigorously. A dropper is provided to count the drops. The suspension must be shaken vigorously before every use. Compliance will be monitored by filling out a diary.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged between 30 and 90 days
* Breast fed exclusively during length of trial
* Diagnosis of infantile colic according to Wessel's criteria i.e paroxysmal fussing in infancy for more than three hours per day, at least three days per week but not treated previously for colics.
* Debut of colic symptoms 6+/-1 days before randomization
* Written informed consent from one or both parents
* Stated availability and reliability throughout the study period.

Exclusion Criteria:

* Major chronic disease
* Gastrointestinal disease
* Administration of antibiotics the week before randomization
* Administration of probiotics two weeks before randomization
* Infants with GI malformation, cystic fibrosis, other genetic diseases
* Participation in other clinical trials.

Ages: 30 Days to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Improvement of colics symptoms | 3 weeks
  improvement of colics symptoms by the oral administration of probiotic VSL#3 drops

SECONDARY OUTCOMES:
Difference in the daily average crying time between end of treatment and baseline. | 3 weeks
  Difference in the daily average crying time, measured with parental diary, between end of treatment and baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Mariella Baldassarre, PhD, Principal Investigator — Policlinico Hospital
Locations (1):
- Dept Of Obstetrics and Neonatology - Section of Neonatology University of Bari Policlinico Hospital, Bari, Italy

REFERENCES:
- [Derived] Baldassarre ME, Di Mauro A, Tafuri S, Rizzo V, Gallone MS, Mastromarino P, Capobianco D, Laghi L, Zhu C, Capozza M, Laforgia N. Effectiveness and Safety of a Probiotic-Mixture for the Treatment of Infantile Colic: A Double-Blind, Randomized, Placebo-Controlled Clinical Trial with Fecal Real-Time PCR and NMR-Based Metabolomics Analysis. Nutrients. 2018 Feb 10;10(2):195. doi: 10.3390/nu10020195. PMID 29439395